CLINICAL TRIAL: NCT04561388
Title: Usefulness of Electrocochleography for the Longitudinal Evaluation of Residual Hearing in Hearing Rehabilitation With Cochlear Implant
Brief Title: Electrocochleography Along Cochlear Implant Auditory Rehabilitation
Acronym: eCochGIC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: patient recruitment problem
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL18_0926
Record Dates: First submitted 2020-09-16; First posted 2020-09-23 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Cochlear Prosthesis Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cochlear implant candidates with measurable residual hearing (Other): Electrocochleography responses to acoustic will be recorded during the cochlear implantation and the 6 first months of use of the cochlear implant.
  A pure tone audiometry will be done prior and after the implantation. Speech audiometry will be done twice after the cochlear implantation.
  Interventions: Procedure: Electrocochleography; Other: Pure Tone Audiometry; Other: Speech audiometry

INTERVENTIONS:
Procedure: Electrocochleography — Electrocochleographic responses will be evoked using different pure tone sounds delivered through an insert placed in the external auditory duct. The responses will be recorded with the electrodes of the cochlear implant connected to a dedicated interface.
  Electrocochleographic responses will be collected continuously during the electrode-array insertion at the implantation surgery using 500Hz pure tone and after suturing with 250, 500, 750 and 1000Hz pure tones. Then, electrocochleographic responses to pure tones from 125 to 8000HZ (according to the subject residual hearing) will be recorded 2 weeks, 1 month, 2 months and 4 months after implantation.
Other: Pure Tone Audiometry — The perception thresholds to 125, 250, 500, 750, 1000, 2000, 4000 and 8000 Hz pure tones will be measured within the month preceding the implantation using the same insert t.
  Pure tone audiometry with the same frequencies will be done 2 weeks, 1, 2 and 4 months after the implantation.
Other: Speech audiometry — The speech perception will be assessed in silence and in noise in free field 1 and 4 months after implantation. The speech perception in silence will be assessed using monosyllabic words 60 dB SPL. Speech in noise will be assessed using an adaptative test with fixed noise level (60 dB SPL).

SUMMARY:
Electrocochleography (eCochG) is an electrophysiological measurement to evaluate the activity of cochlear hair cells in response to acoustic stimulation. This measure thus reflects the functional state of the cochlea and more specifically the neuronal survival.

Whereas in the normal-hearing subject, eCochG collection requires the introduction of a collection electrode in the middle ear, closest to the cochlea, in the cochlear implant subject, eCochG can be collected through the electrodes of the cochlear implant.

Measured during surgery, eCochGs may help optimize the placement of the electrode array within the cochlea and help in the decision to refer the patient to a conventional cochlear implant or, when residual cochlear activity is detected, to an electro-acoustic implant system.

The main objective of this study is to evaluate the usefulness of intra-operative eCochG collections for the optimization of electrode array placement within the cochlea and then for monitoring the residual hearing and its relationship to hearing performance during the first months of rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, male or female, aged 8 to 75 ;
2. Candidates for cochlear implantation with measurable residual hearing?
3. French must be the mother tongue and is (or has been) the language of schooling;
4. No ototoxic or neurotropic drug treatment (epilepsy, behavioral disorders, other neurological impairment);
5. No known cognitive disorders, neurodegenerative disorders (Alzheimer's, Parkinson's, ...), psychiatric pathologies (depression, schizophrenia, eating disorders, ...) or neurodevelopmental disorders (attention deficit disorder with or without hyperactivity, autism spectrum disorder, specific learning disorder);
6. Absence of uncorrected visual problems;
7. Normal ENT examination;
8. Valid membership in a social security system;
9. Non-participation in another study;
10. Absence of exposure to loud noise in the 72 hours preceding the experiments;
11. Written consent to free and informed participation signed by the subject and his/her legal guardians in the case of minors.

Exclusion Criteria:

1. Absence of signature of the informed consent by the adult subject and/or the parents of the minor subject ;
2. Subjects speaking a foreign language at home and/or whose schooling was conducted in a foreign language (except for subjects attending bilingual schools and one of whose parents' usual language is French);
3. Subjects undergoing ototoxic or neurotropic drug treatment (epilepsy, behavioural disorders, other neurological impairment);
4. Subjects suffering from cognitive deficits, neurodegenerative disorders (Alzheimer's, Parkinson's, ...), psychiatric pathologies (depression, schizophrenia, eating disorders, ...) or neurodevelopmental disorders (attention deficit disorder with or without hyperactivity, autism spectrum disorder, specific learning disorder);
5. General state of health incompatible with the protocols;
6. Disability(ies) associated with deafness (deaf-blindness, ...) ;
7. Exposure to intense noise in the 72 hours preceding the experiment.
8. Non-affiliation to a social security system.
9. Pregnant or breastfeeding woman
10. Subjects deprived of liberties

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Change in Electrocochleographic responses | During surgery to 4 month after implantation
  The amplitudes of electrocochleographic responses (in µV) to the selected acoustic pure tones will be collected.

SECONDARY OUTCOMES:
Pure tone thresholds | before implantation, 2 weeks, 1 month, 2 month and 4 month after implantation
  The perception thresholds (in dB HL) of the selected acoustic pure tones will be collected.
  No safety issue
Speech audiometry measurements | 1 month , 4 month
  For the speech audiometry in silence, the percentage of correct recognition of monosyllabic words' list will be collected. For the speech audiometry in noise, the signal noise ratio(s) (in dB) permitting the subject to reach 50% and/or 70% of speech recognition (SRT50 and SRT70) will be estimated.
  No safety issue

CONTACTS AND LOCATIONS:
Overall Officials: Hung THAI VAN, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hopital Edouard Herriot, Lyon, France